CLINICAL TRIAL: NCT02683135
Title: Low-carbohydrate Diet, With or Without Exercise, for Improving Postprandial Glucose Control and Vascular Function in Type 2 Diabetes and Prediabetes.
Brief Title: Lifestyle Control of Postprandial Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: H1501952
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, High-Protein Low-Carbohydrate; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-carbohydrate diet (Active Comparator)
  Interventions: Behavioral: High-carbohydrate diet
- Low-carbohydrate diet (Experimental)
  Interventions: Behavioral: Low-carbohydrate diet
- Low-carbohydrate diet with post-meal walking (Experimental)
  Interventions: Behavioral: Low-carbohydrate diet; Behavioral: Low-carbohydrate diet with post-meal walking

INTERVENTIONS:
Behavioral: High-carbohydrate diet — Participants will engage in 4 days of high-carbohydrate low fat diet as recommended by the Canadian Diabetes Association. The macronutrients content will go as follow: 55% carbohydrate, 25% protein and 20% fat. Breakfast, lunch and dinner will be provided to the participants as part of an isoenergetic diet. Between interventions there will be at least a one-week washout, where participants are encouraged to return to their baseline dietary habits.
  Arms: High-carbohydrate diet
Behavioral: Low-carbohydrate diet — Participants will engage in 4 days of low-carbohydrate high-fat diet. The macronutrients content will go as follow: 10% carbohydrate, 25% protein and 65% fat. Breakfast, lunch and dinner will be provided to the participants as part of an isoenergetic diet. Between interventions there will be at least a one-week washout, where participants are encouraged to return to their baseline dietary habits.
  Arms: Low-carbohydrate diet; Low-carbohydrate diet with post-meal walking
Behavioral: Low-carbohydrate diet with post-meal walking — Participants will follow the same diet as in the low-carbohydrate diet arm but also perform 15 minutes of walking beginning ~15 minutes after breakfast, lunch and dinner. Approximately 70 kcal (individualized) will be added to main meals to account for exercise energy expenditure. Between interventions there will be at least a one-week washout, where participants are encouraged to return to their baseline dietary habits.
  Arms: Low-carbohydrate diet with post-meal walking

SUMMARY:
Large spikes in blood glucose experienced after meals in people with type 2 diabetes are known to damage blood vessels. Low carbohydrate high fat diets and exercise can improve blood glucose control in people with type 2 diabetes but it is unclear how these two strategies interact to affect blood vessel function and inflammation. We will examine how following a short-term low carbohydrate high fat diet (4 days) with or without post-meal walking impacts markers of blood vessel function and inflammation. We will also examine how a single low carbohydrate high fat meal, with or without post-meal walking, impacts blood glucose control and blood vessel function. Findings will help determine the best lifestyle approach for improving cardiovascular health in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes (at least 6 months ago)
* Aged 40-75
* Engaging in 2 or less moderate-to-vigorous exercise bouts per week in the last 3 months
* Ability to understand and communicate in English to interact with the personal trainer

Exclusion Criteria:

* Diagnosed coronary artery disease
* Any contraindications to exercise (e.g., musculoskeletal injury)
* Prior history of cardio- or cerebrovascular disease or myocardial infarction
* Hypertension that is not controlled by medication (systolic blood pressure (BP) >160 mmHg and/or diastolic BP >99 mmHg)
* Change in diabetes medications in the previous 6 months
* Diagnosed with peripheral neuropathy
* Taking exogenous insulin

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Difference in glycemic control assessed by continuous glucose monitoring in low-carbohydrate, low-carbohydrate plus post-meal walking, and high-carbohydrate low-fat arm. | 4-day average glucose levels assessed in each arm.

SECONDARY OUTCOMES:
Change from baseline in circulating inflammatory cytokines after 4 days of intervention. | Fasting measurements taken on day 1 and day 5.
Change from baseline in toll-like receptors 2 and 4 expression on white blood cells after 4 days of intervention. | Fasting measurements taken on day 1 and day 5.
Change from baseline in flow mediated dilation of brachial artery after 4 days of intervention. | Fasting measurements taken on day 1 and day 5.

OTHER OUTCOMES:
Change from baseline in flow-mediated dilation after single breakfast meal on day 1 of the intervention | Baseline and 1, 2, and 3 hours post-breakfast on day 1 in each arm
Change from baseline in plasma glucose after single breakfast meal on day 1 of the intervention | Baseline and 1, 2, and 3 hours post-breakfast on day 1 in each arm
Change from baseline in body weight after a single meal and 4 days of intervention. | Fasting measures on day 1 and day 5.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Little, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No